CLINICAL TRIAL: NCT03698903
Title: Evaluating the Effects of a Sedentary Behavior Reduction Intervention on the Sedentary Time and Blood Pressure of Overweight/Obese Adults
Brief Title: Take a STAND 4 Health: A Sedentary Behavior Reduction Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Responsible Party: Principal Investigator, Chelsea Larsen, Graduate Student, University of South Carolina
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: Pro00079096
Record Dates: First submitted 2018-09-17; First posted 2018-10-09 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Blood Pressure
Keywords: Intervention; Sedentary Behavior; Overweight or obese adults
MeSH Terms: conditions — Sedentary Behavior; Overweight

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Take a STAND 4 Health: Immediate (Experimental): Receives the coaching calls + mHealth intervention first, then receives only the mHealth intervention after the 4 week assessment.
  Interventions: Behavioral: Take a STAND 4 Health
- Take a STAND 4 Health: Delayed (Active Comparator): Will receive no intervention for the first 4 weeks but then after assessment will be provided the opportunity to receive the full coaching calls + mHealth intervention.
  Interventions: Behavioral: Take a STAND 4 Health

INTERVENTIONS:
Behavioral: Take a STAND 4 Health — The 4-week is comprised of several elements, including: (1) an in-person introductory session to acquaint the individuals with all intervention elements, customize to their preferences and describe the mHealth component of the intervention; (2) a website that will provide individualized feedback over time on the participant's scheduled breaks, sedentary time reduction, and sedentary patterns; (3) texts to serve as prompts and alert the participant to stand or move, with a goal of a 60 minute reduction per day, which are customized to the individual's schedule, personal preference and sedentary profile; and (4) two coaching phone calls to trouble shoot and problem solve implementation of the intervention.

SUMMARY:
There is emerging evidence that an excessive amount of sitting is linked with an increased risk of negative health outcomes independent of an individual's physical activity levels. This is concerning considering data indicate Americans spend over half of the waking day engaged in sedentary activities, and that individuals who are overweight or obese and/or have a chronic disease such as hypertension are likely to have an even higher level of sedentary behavior. A limited number of experimental studies have looked at the effects of reducing sitting time on blood pressure and have shown promise. However, these studies lasted for only a day, so it is unclear how reducing sedentary time may influence blood pressure over a longer duration. The purpose of this study is to look the relationships between the amount of time a person spends sitting and their blood pressure and examine whether decreasing sedentary behavior helps improve blood pressure. The study employs the use of coaching calls and a mobile health (mHealth) intervention to reduce the sedentary behavior of participants through strategies such as prompting, feedback, and counseling.

DETAILED DESCRIPTION:
The purpose of this study is to determine the effect of a 4-week sedentary behavior reduction intervention on objectively measured sedentary behavior of overweight or obese adults. The proposed study is a pilot, proof-of-concept randomized controlled trial that will randomize participants to either the 1) Immediate Intervention group, which will receive coaching calls + a mHealth intervention for the first four weeks of the study and then will receive only the mHealth intervention for the remaining 4 weeks or the 2) Delayed Intervention Control group, which will act as an assessment-only condition for the first 4 weeks and then will receive the coaching calls + mHealth intervention for 4-weeks. This design has two phases: Phase 1, which is a randomized controlled feasibility pilot and the primary study focus, followed by Phase 2, which is an exploratory phase, allowing replication of the intervention (in the Delayed Intervention Control group) and extended follow-up (in the Immediate Intervention group).

The study outcomes to be investigated in Phase 1 include:

* 1) the change in total % sedentary time from baseline to the 4-week assessment, comparing the average proportion of objectively-measured time spent sitting during the waking day across the previous week in the Immediate Intervention group (which will have received the 4-week coaching calls + mHealth sedentary behavior reduction intervention) with the average proportion of objectively-measured waking sedentary time across the previous week in the Delayed Intervention Control group (which will have received assessment only during this period).
* 2) the change in blood pressure, comparing the Immediate Intervention group (which will have received the 4-week coaching calls + mHealth sedentary behavior reduction intervention) with the Delayed Intervention Control group (which will have received assessment only during this period).
* 3) Process data on participant recruitment to the study, and, among those randomized to the Immediate intervention, engagement with the intervention (e.g., response rates to the texts, completion of intervention phone calls, etc.), and participant evaluation of the intervention.

The study outcomes to be investigated in Phase 2 include:

* 1) Objectively measured sedentary behavior in the Immediate Intervention group 4 weeks post-treatment (i.e. at 8-week assessment), allowing quantification of maintenance of sedentary behavior reduction following the termination of coaching calls.
* 2) Objectively-measured sedentary behavior and blood pressure at 8 weeks post randomization in the Delayed Intervention Control group (i.e. following implementation of the 4-week coaching calls+ mHealth intervention), allowing assessment of whether intervention effects are reproducible.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years or older
* Having a BMI between 25 and 50 kg/m2
* Owning a smartphone that is accessible during the day
* Living or working within 30 miles of University of South Carolina (USC)
* Willing to wear the activPAL for baseline assessment
* An average self-reported sedentary time of at least 7 hours over the past 7 days
* Willing to be randomized to either group

Exclusion Criteria:

* Inability to walk without assistance
* Recent use of psychotropic medications or treatment for psychological issues, with the exception of anxiety and depression
* Current treatment for cancer or other serious medical conditions such as renal failure
* Injury or illness that prohibits standing or walking
* Pregnant or gave birth within the last 6 months
* Does not live or work within 30 miles of USC
* Currently enrolled in a weight loss, physical activity, or stress management program
* A known vacation or a major alteration in their normal schedule in the next 4 months
* Unwilling to wear the accelerometer for 7 days at any assessment period or had an adverse reaction to wearing the accelerometer during baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-11-15 (Actual)

PRIMARY OUTCOMES:
Change in percent time spent sedentary | Baseline, 4 weeks, 8 weeks
  activPAL device

SECONDARY OUTCOMES:
Blood pressure | Baseline, 1 week, 4 weeks, 8 weeks
  Automated blood pressure machine
Percent time spent in light physical activity | Baseline, 4 weeks, 8 weeks
  activPAL device
Percent time spent in moderate-to-vigorous physical activity | Baseline, 4 weeks, 8 weeks
  activPAL device
Self-reported sedentary behavior | Baseline, 1 week, 4 weeks, 8 weeks
  The Sedentary Behavior Questionnaire is assesses domain specific sedentary time on both a weekday and weekend. The scale ranges from "none" to "6 or more hours" for each sedentary activity, with a higher value indicating a higher amount of sedentary time. All responses are summed and the value is the individuals sedentary time.
Self-reported physical activity | Baseline, 4 weeks, 8 weeks
  The International Physical Activity Questionnaire- Short form measures the frequency (0-7 days) and amount of time (number of hours and minutes) an individual spends in vigorous intensity physical activity, moderate intensity physical activity, and walking. The total number of metabolic equivalent (MET) minutes per week are calculated from these responses. The survey also assess an individuals total sedentary time on a weekday.
Waist circumference | Baseline, 1 week, 4 weeks, 8 weeks
  Gulick tape
Weight | Baseline, 1 week, 4 weeks, 8 weeks
  Calibrated Tanita body weight scale that measures weight in both pounds and kilograms.
Height | Baseline
  Stadiometer
Treatment Satisfaction | 4 weeks, 8 weeks
  Survey

CONTACTS AND LOCATIONS:
Overall Officials: Chelsea Larsen, MPH, Principal Investigator — University of South Carolina
Locations (1):
- University of South Carolina, Columbia, South Carolina, United States